CLINICAL TRIAL: NCT07405372
Title: Construction and Application of an IDH Mutation-Targeted PET/MRI Imaging Framework for Precision Diagnosis of Gliomas
Status: Recruiting | Type: Observational
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Xiao Chen, Director of Nuclear Medicine Department, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Other Study IDs: 2025460
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Glioma
Keywords: Glioma, IDH, PET/MRI
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — histopathological findings obtained from biopsy or resected surgical specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Targeted IDH PET/MRI — Patients with clinical suspected gliomas will receive the targeted IDH PET/MRI.

SUMMARY:
Glioma is the most common primary intracranial tumor in adults, with high-grade gliomas accounting for more than 50% of all gliomas and having the highest mortality rate. The molecular characteristics of gliomas are closely associated with the selection of treatment regimens, therapeutic efficacy, and patient prognosis. Mutations in isocitrate dehydrogenase (IDH) are an important diagnostic marker for diffuse gliomas and a key component in distinguishing and defining glioma subtypes. Furthermore, the advent of IDH-targeting inhibitors has brought hope to patients with IDH-mutant gliomas. Therefore, accurately assessing the IDH mutation status of gliomas is a prerequisite and key to precision diagnosis, targeted therapy, and prognostic evaluation. This study explores the application value of targeted IDH PET/MRI imaging in glioma subtype diagnosis, tumor grading, and prognostic evaluation. It aims to establish a non-invasive in vivo tracing technology platform and evaluation system for accurately assessing glioma IDH mutation status, subtype diagnosis, and prognostic evaluation. This will provide a basis for the precise diagnosis of gliomas, the selection of targeted treatment regimens, and prognostic assessment, and promote future research and development of therapeutic drugs using labeled therapeutic radionuclides.

DETAILED DESCRIPTION:
1. Clinical and biological data: The records include all patients' general clinical information, disease course, and other imaging findings.
2. PET image analysis: Record and assess lesion location, size, maximum standardized uptake (SUVmax), and target-to-species ratio (TBR), where the TBR value is calculated by dividing the SUVmax of the lesion by the background SUVmean.
3. Pathological analysis: Hematoxylin and eosin staining and immunohistochemical analyses will be performed. Immunohistochemical analysis will be used to investigate the status of isocitrate dehydrogenase (IDH).

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age at the time of consent;
* Patients with suspected, newly diagnosed, or previously treated gliomas;
* Provided written informed consent authorisation before participating in the study.

Exclusion Criteria:

* Pregnancy or lactation;
* MRI contraindications, not limited to cardiac implantable electronic devices and claustrophobia;
* Participants with radiation exposure exceeding 50 mSv in the past year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects the investigators selected are adults who are not restricted by gender.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic efficacy, survival analysis | Completed within half year after end of the study
  sensitivity, specificity, accuracy, positive and negative predictive values, ROC curve analysis,

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Chen, Principal Investigator — Daping Hospital, Army Medical University
Locations (1):
- Department of Nuclear Medicine, Daping Hospital of Army Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaiser L, Quach S, Zounek AJ, Wiestler B, Zatcepin A, Holzgreve A, Bollenbacher A, Bartos LM, Ruf VC, Boning G, Thon N, Herms J, Riemenschneider MJ, Stocklein S, Brendel M, Rupprecht R, Tonn JC, Bartenstein P, von Baumgarten L, Ziegler S, Albert NL. Enhancing predictability of IDH mutation status in glioma patients at initial diagnosis: a comparative analysis of radiomics from MRI, [18F]FET PET, and TSPO PET. Eur J Nucl Med Mol Imaging. 2024 Jul;51(8):2371-2381. doi: 10.1007/s00259-024-06654-5. Epub 2024 Feb 24. PMID 38396261